CLINICAL TRIAL: NCT06036498
Title: Evaluation of Cerebral Blood Flow and Cerebral Oxygenation With Transcranial Doppler and NIRS in Laparoscopic Cholecystectomy Cases
Acronym: NIRS L/C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Kadir Bugra Basaran, Medical Doctor, Research Assistant at Department of Anesthesiology and Reanimation, Uludag University
Other Study IDs: Bursa Uludag Universitesi
Record Dates: First submitted 2023-08-30; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Cerebral Hypoperfusion; Cerebral Occlusion; Cholecystitis; Gallstone; Cholecystitis/Cholelithiasis
Keywords: Near Infra-Red Spectrophotometry; Cerebral Oxygenisation; Transcranial Doppler Ultrasonography (TCD); Laparoscopic Surgery
MeSH Terms: conditions — Cerebrovascular Disorders; Cholecystitis; Gallstones; Cholelithiasis | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- Preoperative Assessment of Trail Group
  Interventions: Device: Near Infrared Spectrophotometry Device, Transcranial Doppler Ultrasonography
- Post-Anaesthetic Induction Assessment of Trial Groups
  Interventions: Device: Near Infrared Spectrophotometry Device, Transcranial Doppler Ultrasonography
- After Pneumoperitoneum Assessment of Trial Groups
  Interventions: Device: Near Infrared Spectrophotometry Device, Transcranial Doppler Ultrasonography
- Within Head-up Tilt Position Assessment of Trial Groups
  Interventions: Device: Near Infrared Spectrophotometry Device, Transcranial Doppler Ultrasonography
- Neuralized Position Assessment of Trial Groups
  Interventions: Device: Near Infrared Spectrophotometry Device, Transcranial Doppler Ultrasonography
- Within Deflation of Abdomen Assessment of Trial Groups
  Interventions: Device: Near Infrared Spectrophotometry Device, Transcranial Doppler Ultrasonography
- Awaking Period from Anaesthesia Assessment of Trial Groups
  Interventions: Device: Near Infrared Spectrophotometry Device, Transcranial Doppler Ultrasonography

INTERVENTIONS:
Device: Near Infrared Spectrophotometry Device, Transcranial Doppler Ultrasonography — We will get signals from the NIRS probes which are positioned bitemporal region of forehead in same time testing intracranial blood flow via TCD device.
  Other Names: NIRS; iNVOS Spectrophotometry

SUMMARY:
The goal of this clinical trial is to test intracranial blood flow and cerebral oxygenisation changes in patients who have pneumoperitoneum in laparoscopic cholecystectomy procedure.

The main questions aim to answer are:

* How does pneumoperitoneum in laparoscopic cholecystectomy procedure changes blod flow in patients?
* Are there any differences between Near-Red spectroscopy and transcranial doppler ultrasonography assesment?

Participants will be diagnosed with using NIRS probes and Doppler ultrasonography probes if any changes in surgical procedure.

Researchers will compare NIRS and TCD detection outcomes to see if there is any differences.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is the gold standard treatment method for benign gallbladder stones. The required pneumoperitoneum for the operation leads to hemodynamic and metabolic changes in patients. Prolonged complicated laparoscopic surgeries also pose an additional risk factor for neurological complications.

Cerebral circulation occurs within a closed environment enclosed by the skull. This environment includes brain tissue, blood volume, and cerebrospinal fluid. Cerebral blood pressure arises from the difference between arterial blood pressure and intracranial pressure. Due to carbondioxide insufflation in laparoscopic surgery, caused by pneumoperitoneum creation, intra-abdominal carbondioxide is rapidly absorbed through the peritoneal membrane and enters the bloodstream.

Carbonic acid formed by the carbonic anhydrase enzyme in the plasma leads to respiratory acidosis. The resulting respiratory acidosis triggers peripheral and central vasodilation to ensure oxygenation and gas exchange, causing a rightward shift in the hemoglobin curve. Hypercarbia's impact on cells and the effect of cellular acidosis lead to local tissue edema. All of these factors contribute to changes in transcranial pressure. An increase in intracranial pressure can result in impaired cerebral perfusion.

Transcranial Doppler (TCD) is a reliable tool for imaging intracranial pressure due to its affordability, non-invasiveness, repeatability at the bedside, and real-time data provision during acute situations. Transcranial Doppler ultrasonography (TCD) can better display flow velocity waveforms, flow direction, intraparenchymal flow velocity, and density compared to other diagnostic tests. Changes in waveforms detected by TCD allow tracking changes in intracranial pressure. However, assessing tissue oxygenation solely with transcranial Doppler ultrasonography is not feasible.

Near-Infrared Spectroscopy (NIRS) can play an effective role in showing tissue oxygen perfusion for this purpose. NIRS imaging, similar to pulse oximetry, utilizes infrared light between 650 and 1000 nm to measure oxyhemoglobin levels in tissues and capillaries. Its non-invasiveness, ease of tolerance by the patient, and ability to quickly detect sudden drops in oxygen levels in tissues make it reliable.

In this study, Researchers aimed at implementing in patients planned for laparoscopic cholecystectomy, intend to use TCD and NIRS protocols to detect changes in intracranial blood flow and cerebral tissue oxygenation during the preoperative, intraoperative, and postoperative periods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiology (ASA) 1-3 classification,
* Both male and female patients between the ages of 18 to 65,
* Patients scheduled for elective laparoscopic cholecystectomy.

Exclusion Criteria:

* American Society of Anesthesiology (ASA) 4 and above patient groups,
* Patients aged under 18 and over 65,
* Patients with a history of known previous cerebrovascular accident (CVA),
* Patients with follow-up due to Cerebrovascular Ischemic Brain Attack Syndrome (CIBAS),
* Patients diagnosed with Carotid Stenosis,
* Patients diagnosed with peripheral and central vascular diseases,
* Patients with general debilitation and extreme senility,
* Cases that require conversion to laparotomy during the intraoperative period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who has;
  * Cholelithiasis,
  * Gallbladder Stones,
  * Diagnosed with acute cholecystitis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-26 (Estimated)

PRIMARY OUTCOMES:
Detecting Cerebral Blood Flow Changes at Pneumoperitoneum Time via New Assessment Methods | Perioperative Time in Laparoscopic Cholecystectomy Surgery Procedures
  In this study, aimed at patients scheduled for laparoscopic cholecystectomy, Researchers intend to utilize transcranial doppler ultrasonography to detect changes in intracranial blood flow changes during the preoperative, intraoperative, and postoperative periods.
Detecting Cerebral Tissue Oxygenisation Changes at Pneumoperitoneum Time via New Assessment Methods | Perioperative Time in Laparoscopic Cholecystectomy Surgery Procedures
  In this study, aimed at patients scheduled for laparoscopic cholecystectomy, Researchers intend to utilize Near Infrared spectrophotometry methods to detect oxygenisation changes in cerebral hemispheres during the preoperative, intraoperative, and postoperative periods.

OTHER OUTCOMES:
Detecting any difference between Near Infrared Spectrophotomery and Transcranial Doppler | Perioperative Time in Laparoscopic Cholecystectomy Surgery Procedures
  Researchers will compete Near Infrared spectrophotometry and transcranial doppler ultrasonography methods in cerebral hemodynamics in perioperative process in laparoscopic cholecystectomy patients.

CONTACTS AND LOCATIONS:
Overall Officials: Kadir Bugra Basaran, Study Chair — Uludag University
Locations (1):
- Bursa Uludag University, Faculty of Medicine, Department of Anesthesiology and Reanimation, Bursa, Nilufer, Turkey (Türkiye)